CLINICAL TRIAL: NCT04011397
Title: Feasibility of Procedures for a Pragmatic Randomized Controlled Trial of Reduced Exertion, High-intensity Interval Training (REHIT) With Non-diabetic Hyperglycaemia Patients
Brief Title: Feasibility of REHIT in NDH Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Huddersfield (Other)
Responsible Party: Principal Investigator, Matthew Haines, Principal Investigator, University of Huddersfield
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UHuddersfield
Record Dates: First submitted 2019-06-26; First posted 2019-07-08 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Diabetes; Physical Activity
Keywords: Diabetes; Exercise; Feasibility; HbA1c; Interval training
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Exercise intervention (reduced-exertion, high-intensity interval training) alongside normal treatment. [low recruitment prohibited control arm]
  Interventions: Other: Exercise intervention; Behavioral: Usual care

INTERVENTIONS:
Other: Exercise intervention — Exercise intervention (reduced-exertion, high-intensity interval training) delivered within an NHS setting. Consisted 10 min of cycle ergometry (inclusive of warm-up and cool down) including very brief maximal cycle sprints.
Behavioral: Usual care — Members of a multi-disciplinary team including a consultant, diabetes specialist nurse, clinical psychologist, physiotherapist, and dietician worked together to promote patient self-management. Care was tailored to the specific circumstances of each patient after initial assessment and focussed on weight management, dietary education, behavioural therapy, and supported pharmacotherapy initiation as appropriate.

SUMMARY:
The aim of this feasibility study was to describe and report data relevant to the acceptability of an exercise intervention (reduced-exertion, high-intensity interval training) in non-diabetic hyperglycaemia patients delivered in a National Health Service setting.

DETAILED DESCRIPTION:
Background Physical activity and exercise interventions to improve health frequently bring about intended effects under ideal circumstances but fail to demonstrate effectiveness when translated to demonstrable benefits in real-world contexts. The aim of this feasibility study was to describe and report data relevant to the acceptability of an exercise intervention (reduced-exertion, high-intensity interval training) in non-diabetic hyperglycaemia (NDH) patients delivered in a National Health Service (NHS) setting.

Individuals with NDH are an intermediary group of patients whose blood glucose levels are higher than normal but not high enough to be diagnosed as diabetic. Such hyperglycaemic blood glucose excursions in 'pre-diabetic' states contribute to the development of macro- and micro-vascular disease risk and increases the risk of developing overt type 2 diabetes. Interventions - such as increased physical activity - for individuals who are diagnostically considered to have NDH are high priority, as they provide a substantial opportunity for preventing future burden of diabetes on patients, the NHS, and the economy.

Evidence supporting the efficacy of exercise and physical activity as preventative or therapeutic treatments for a range of chronic diseases, including obesity and diabetes, is incontrovertible. However, exercise adherence is considered a significant issue. The most commonly cited barrier to undertaking physical activity is perceived 'lack of time'. Consequently, there has been a recent interest in high-intensity interval training (HIT) which is characterised by brief periods of repeated very high-intensity exercise interspersed with longer periods of recovery. More recently attempts have been made to modify HIT to make it more time-efficient and tolerable. This approach is known as reduced-exertion, high-intensity interval training (REHIT). In this study, issues of acceptability and feasibility were considered when implementing a REHIT intervention into usual care within an NHS setting.

Methods The purpose was to assess whether it would be appropriate to progress to a larger-scale pragmatic trial, and to optimise the design and conduct of any such trial. The intention was to recruit 40 participants from a single centre (specialist diabesity centre). Patients were eligible to take part if they were diagnostically defined as non-diabetic hyperglycaemic based on a glycated haemoglobin value of 42-46 mmol·mol. Methodological issues were used to analyse problems that arose.

ELIGIBILITY:
Inclusion Criteria:

* Accessing the NHS Trust Weight Management Service (Specialist Diabesity Clinic)
* Aged between 18 and 65 years (inclusive)
* Diagnosed as NDH (using standard criteria)
* Male or female
* Any ethnicity
* Not currently partaking in a new structured exercise intervention
* Considered low or medium risk for exercise using standard risk stratification [37]

Exclusion Criteria:

* < 18 years and ≥ 66 years
* Currently partaking in a new structured exercise intervention
* Euglycaemic
* Diagnosed with type 1 or type 2 diabetes; taking insulin; history of end stage liver or kidney disease, neuropathy or retinopathy; has hypertension that cannot be controlled by standard medication; has cardiovascular disease, or another contraindication to exercise
* Considered high risk for exercise using standard risk stratification [37]
* Unable to adequately understand verbal explanations and written information given in English (there were no funds available for translation services)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of patients screened and considered eligible to take part in the study | 4-weeks
  Defined as the number of patients who had contact with the recruitment team and who were assessed for eligibility using inclusion and exclusion criteria.
Reporting of adverse events | From first exposure to intervention to last (approx. 6-weeks)
  An adverse event was defined as any untoward occurrence that happened during the conduct of the study.
Intervention adherence | From first exposure to intervention to last (approx. 6-weeks)
  Intervention adherence was calculated by summing the total number of participants and the target number of REHIT sessions (15 per participant) and comparing this against the actual completed sessions.
Change in affective valence (pleasure-displeasure) | Change from first exposure to intervention to last (approx. 6 weeks)
  Pre-validated 'Feeling Scale' questionnaire which measure pleasure/displeasure responses during exercise. This is a single-item, 11-point, bipolar scale and ranges from - 5 'very bad' to + 5 'very good', with anchors designated for 0 (neutral) and all odd integers in-between. Lower scores are considered to be a worse outcome.
Change in perceived exertion | Change from first exposure to intervention to last (approx. 6 weeks)
  Pre-validated 'Rating of Perceived Exertion' questionnaire which measures perceived effort during exercise. This is a 15-point scale and ranges from 6 'no exertion' to 20 'maximal exertion' with anchors designated for all the odd integers in-between. A higher score is considered a worse outcome.
Change in enjoyment | Change from first exposure to intervention to last (approx. 6 weeks)
  Pre-validated 'Exercise Enjoyment Scale' (ESS) which measures enjoyment associated with exercise. This is a single-item, 7-point scale. Anchors are given at every integer, ranging from 1 'not at all' to 7 'extremely'. A lower score is a worse outcome.

SECONDARY OUTCOMES:
Change in peak oxygen uptake (fitness test) | Change from baseline peak oxygen uptake at approx. 6-weeks
  Progressive cycle test to measure cardiovascular fitness (using gas analysis)
Change in HBA1c (blood test) | Change from baseline HbA1c at approx. 6-weeks
  Widely used measure of blood glucose control
Change in body composition | Change from baseline body composition at approx. 6-weeks
  Fat mass and fat-free mass estimated via bioelectrical impedance analysis
Change in systolic and diastolic blood pressure | Change from baseline systolic and diastolic blood pressure at approx. 6-weeks
  Measured via automated digital blood pressure monitor

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Haines, Principal Investigator — University of Huddersfield

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Haines M. Feasibility of procedures for a randomised pilot study of reduced exertion, high-intensity interval training (REHIT) with non-diabetic hyperglycaemia patients. Pilot Feasibility Stud. 2020 Feb 19;6:28. doi: 10.1186/s40814-020-00571-8. eCollection 2020. PMID 32099663